CLINICAL TRIAL: NCT05348954
Title: Determining the Effects of Sexual Health Education and Counseling Given to Women in the Postpartum Period Based on the EX-PLISSIT Model on Sexual Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Nergiz Eryilmaz, Principal Investigator, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: study1
Record Dates: First submitted 2022-02-14; First posted 2022-04-27 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Sexuality; Nurse's Role; Postpartum Disorder
MeSH Terms: conditions — Sexuality; Puerperal Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sexual dysfunction of women (Experimental): Sexual dysfunction of women
  Interventions: Other: EX-PLISSIT MODEL
- Quality of sexual life (Experimental): Quality of sexual life
  Interventions: Other: EX-PLISSIT MODEL

INTERVENTIONS:
Other: EX-PLISSIT MODEL — The content of the program will include information about the anatomy and physiology of the male-female reproductive system, sexuality and sexual cycle physiology, factors affecting sexuality, postpartum changes, hormonal changes, breastfeeding and their effects on sexuality, and methods of contraception.

SUMMARY:
The aim of this study will be to determine the effect of the sexual health education and counseling program, which is given to women in the postpartum period based on the Ex-PLISSIT model, on women's sexual life, including sexual function, sexual distress and sexual life quality.

DETAILED DESCRIPTION:
The study is a multicenter, parallel randomized controlled experimental study with block randomization.For the determination of the working groups, the researcher; will give general information about the research to women who have applied to the family health center and meet the inclusion criteria in the postpartum period of 10 weeks-6 months and agree to participate, and will receive their written and verbal consent for participation.

ELIGIBILITY:
Inclusion Criteria:

* Being primiparous
* Having given birth at 38-42 weeks of gestation,
* Having a single birth,
* Not experiencing any postpartum complications
* The time elapsed from birth is between 10 weeks and 6 months
* Being sexually active
* Having a spouse/partner
* Having a smartphone or computer with a camera
* Being at least literate

Exclusion Criteria:

* A previous sexual function of the woman herself or her husband.
* Having a chronic disease that she expresses herself (such as cardiovascular disease, hypertension, etc.)
* Having a health problem that requires the baby to be hospitalized
* Having received sexual education/counselling
* Spouse or self-diagnosed mental problem
* Having a diagnosis that will affect sexual function or body image, such as mastectomy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The population of the study will be composed of women who are registered to family health centers determined by randomization in Karaman city center and who are in the 10 weeks-6 months postpartum period.
Enrollment: 88 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-06-02 (Estimated)

PRIMARY OUTCOMES:
EX-PLISSIT Model | EX-PLISSIT Model will be conducted to participants one weeks later after the first session
  The content of the program will include information about the anatomy and physiology of the male-female reproductive system, sexuality and sexual cycle physiology, factors affecting sexuality, postpartum changes, hormonal changes, breastfeeding and their effects on sexuality, and methods of contraception.
THE FEMALE SEXUAL DISTRESS SCALE-REVISED | They will get an sexual health education and then their sexual disstress will be measured 4 weeks later
  Measuring sex-related personal distress for women
SEXUAL QUALITY OF LIFE SCALE-FEMALE | They will get an sexual health education and then their sexual quality of life will be measured 4 weeks later
  This scale measures the quality of sex life.

CONTACTS AND LOCATIONS:
Locations (1):
- Karaman Halk Sağlığı Müdürlüğü, Karaman, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No